CLINICAL TRIAL: NCT05226897
Title: A Multicenter, Double-blind, Placebo-controlled, Randomized, Parallel Group, Phase 3 Study to Evaluate the Efficacy and Safety of YYC405-T Added to Metformin and Dapagliflozin in Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control With the Combination of Metformin and Dapagliflozin
Brief Title: Clinical Trial to Assess the Efficacy and Safety of YYC405 in Type 2 Diabetes Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yooyoung Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YYPCT_YYC405_301
Record Dates: First submitted 2022-01-17; First posted 2022-02-07 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: a Multicenter, Double-blind, Placebo-controlled, Randomized, Parallel group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental): Take YYC405-T and Metformin≥1000mg, Dapagliflozin 10mg
  Interventions: Drug: YYC405-T; Drug: Metformin≥1000mg; Drug: Dapagliflozin 10mg
- Placebo control (Placebo Comparator): Take YYC405-T Placebo and Metformin≥1000mg, Dapagliflozin 10mg
  Interventions: Drug: Metformin≥1000mg; Drug: Dapagliflozin 10mg; Drug: YYC405-T placebo

INTERVENTIONS:
Drug: YYC405-T — Subjects take the investigational products once a day for 24 weeks.
  Arms: Test
Drug: Metformin≥1000mg — Subjects take the investigational products once a day for 24 weeks.
Drug: Dapagliflozin 10mg — Subjects take the investigational products once a day for 24 weeks.
Drug: YYC405-T placebo — Microcrystalline cellulose, Subjects take the investigational products once a day for 24 weeks.
  Arms: Placebo control

SUMMARY:
Phase 3 study to assess the Efficacy and Safety of YYC405 in Type 2 Diabetes Patients

DETAILED DESCRIPTION:
Phase 3 study to assess the Efficacy and Safety of YYC405-T when added to Metformin and Dapagliflozin combination therapy in patients with type 2 diabetes mellitus who have inadequate glycemic control

ELIGIBILITY:
Inclusion Criteria:

* Patient who contsent to participate in this tiral by written informed consent form
* A man or woman over 20 years old
* Type 2 Diabetes patients

Exclusion Criteria:

* Patients with severe renal impairment, end-stage renal disease or on dialysis
* Type 1 diabetes patients
* Patients with a history of acute or chronic target acidosis, including lactic acidosis and diabetic ketoacidosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-06-26 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Baseline, 24 weeks
  Change from baseline in Glycosylated Hemoglobin (HbA1c)

SECONDARY OUTCOMES:
HbA1c | Baseline, 12weeks
  Change from baseline in Glycosylated Hemoglobin (HbA1c)
FPG, Fasting insulin | Baseline, 12weeks, 24weeks
  Change from baseline in Fasing plasma glucose and Fasting insulin
C-peptide | Baseline, 12weeks, 24weeks
  Change from baseline in C-peptide

CONTACTS AND LOCATIONS:
Overall Officials: Sungrae Kim, MD, Ph.D, Study Chair — Bucheon St Mary Hospital
Locations (1):
- The Catholic University of Korea(Bucheon St. Mary's Hospital), Bucheon-si, South Korea

IPD SHARING:
Plan to Share IPD: Undecided